CLINICAL TRIAL: NCT01756261
Title: Special Drug Use Investigation of EYLEA for Quality of Life
Brief Title: EYLEA [AMD-QOL(Age-Related Macular Degeneration-Quality of Life)] Post-marketing Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 16656; EYL-AMD-QOL (Other: company internal)
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Macular Degeneration
Keywords: EYLEA; Age-Related Macular Degeneration; QOL
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Patients treated with EYLEA under practical manner for AMD.

SUMMARY:
The objective of this survey is to evaluate effectiveness of EYLEA on Quality of Life (QOL). The QOL is evaluated by using Japanese version (v.1.4 - interviewer administered format) of National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) and compared at baseline and at the 6 and 12 months after start of EYLEA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been determined to start EYLEA treatment
* Patients who are registered to Special drug use investigation of EYLEA for AMD(Trial Number 15858)
* Patients who have agreed with the patient informed consent

Exclusion Criteria:

* Patients who have already received EYLEA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with subfoveal choroidal neovascular age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2012-12-26 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Changes in mean NEI-VFQ-25 overall scores of patients after the first intravitreal(ITV) injection of EYLEA | From baseline to 6 and 12 months

SECONDARY OUTCOMES:
Changes in mean NEI-VFQ-25 subscale scores of patients after the first ITV injection of EYLEA | From baseline to 6 and 12 months
Changes in mean NEI-VFQ-25 overall scores after the first ITV injection of EYLEA in subpopulations of patient background characteristics and status of EYLEA treatments, ie. Frequency, visual acuity, etc | From baseline to 6 and 12 months
Changes in mean NEI-VFQ-25 subscale scores after the first ITV injection of EYLEA in subpopulations of patient background characteristics and status of EYLEA treatments, ie. Frequency, visual acuity, etc | From baseline to 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan